CLINICAL TRIAL: NCT06833983
Title: A Single-arm, Open-label, Multicenter Study Evaluating the Efficacy and Safety of GS1191-0445 Injection as a Single Dose in Chinese Subjects With Hemophilia A
Brief Title: To Evaluate the Clinical Study of GS1191-0445 Injection in the Treatment of Hemophilia A
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gritgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS1191-0445-GTHA-CN02
Record Dates: First submitted 2025-01-28; First posted 2025-02-19 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-09

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3E12 vg/kg (Experimental)
  Interventions: Drug: GS1191-0445 injection

INTERVENTIONS:
Drug: GS1191-0445 injection — A single intravenous administration of GS1191-0445 injection at a dose of 3E12 vg/kg

SUMMARY:
This study is a single-arm, open-label, multicenter study evaluating the efficacy and safety of GS1191-0445 injection as a single dose in Chinese subjects with hemophilia A.

GS1191-0445 is an AAV8-based gene therapy vector designed to express B-domain deleted human factor VIII (FVIII) under the regulation of a human liver-specific promoter. Following a single intravenous administration, AAV8 targets hepatocytes and facilitates the specific expression and secretion of FVIII into the bloodstream.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the purpose and risks of the study and provide informed consent in accordance with national and local privacy laws:
2. Subject must be male, aged >18 years old at the time of signing informed consent, and ≤65 years old:
3. Participants with confirmed hemophilia A in their pre-admission history and based on clinical laboratory examination ;
4. Subjects had used FVIII products for at least 150 exposure days (ED) before enrollment;
5. Subject has no prior history of FVIII inhibitors;
6. Subjects agree to use a reliable barrier contraceptive method from the date of signing the informed consent
7. Subject is willing and able to follow planned visits, treatment plans, and other study procedures.

Exclusion Criteria:

1. The subject has any hemorrhagic disorder not related to hemophilia A,
2. Abnormal liver function test results of subjects during screening.
3. Abnormal laboratory examination of subjects during screening
4. The subject has acute or chronic hepatitis B virus (HBV) infection or chronic hepatitis C virus (HCV) infection; Or are receiving antiviral treatment for hepatitis B and C;
5. Active systemic immune disease.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Annualized Bleeding Rate (ABR) | Weeks 3 to 52 after infusion
  To evaluate the efficacy of a single intravenous administration of GS1191-0445 in subjects with hemophilia A

SECONDARY OUTCOMES:
Incidence of adverse events (AE) | Within 52 weeks after infusion
  The incidence of adverse events (AE) within 52 weeks after GS1191-0445 infusion, including serious adverse events (SAE) and adverse events of special concern (AESI)
Immunogenic response of AAV8 capsid protein and vector derived FVIII within 52 weeks after GS1191-0445 infusion | Within 52 weeks after infusion
  Evaluate the safety of a single intravenous infusion of GS1191-0445 injection in hemophilia A subjects
Evaluate the long-term efficacy of GS1191-0445 injection after intravenous infusion for 2-5 years | 2-5 years after infusion
  Evaluate the changes in annualized bleeding rate (ABR) and FVIII activity from baseline during the 2nd to 5th year after GS1191-0445 injection

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - First Hospital of Lanzhou University, Lanzhou, Gansu
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - North China University of Science and Technology Affiliated Hospital, Tangshan, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality
  - The second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No